CLINICAL TRIAL: NCT03489174
Title: Routine Pregnancy Screening for Women on Opioid Substitution Therapy: A Randomized Controlled Trial
Brief Title: Routine Pregnancy Screening for Women on Opioid Substitution Therapy
Acronym: PREG-O
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit sufficient participants to complete study intervention
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: PREG-O
Record Dates: First submitted 2018-03-05; First posted 2018-04-05 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Substance Use Disorders; Prenatal Care; Pregnancy Outcome
Keywords: Opioid Substitution Therapy; Pregnancy Tests
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either standard practice or monthly pregnancy screening.
Who Masked: Participant, Investigator
Masking Description: Participants will not know if they are assigned to the intervention or control group. Their weekly urine test that is collected by the opioid substitution therapy clinic will be tested monthly for pregnancy. Pregnancy will then be reported to the patient's attending physician on the day of testing, who would then communicate the result to the patient. The physician will continue with standard pregnancy care. The investigators will remain blind throughout data analysis and will not know if the pregnancy was discovered via monthly testing or standard practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monthly Pregnancy Screening (Experimental): Patients at the Hamilton Clinic present to the clinic most often on a weekly basis to provide a urine sample for urine drug screening and to meet with their MRP. This same urine sample will be tested for pregnancy in the intervention group once per month. Resulting positive test results will be reported to the patient through their attending physician on the day of testing.
  Interventions: Other: Monthly Pregnancy Screening
- Usual Care (Active Comparator): Participants in the control group will not receive study-initiated urine pregnancy testing but will receive usual care, which may include pregnancy testing based on patient request or clinical judgement.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Monthly Pregnancy Screening — Pregnancy test will be administered once per month during weekly urine testing for drug levels.
  Arms: Monthly Pregnancy Screening
Other: Usual Care — Usual care.
  Arms: Usual Care

SUMMARY:
Women who take opioid substitution therapy have higher rates of unintended pregnancy, more pregnancies, and a higher risk of pregnancy complications than the general population. Current practice is to test for pregnancy only at patient request or if the clinician suspects pregnancy. This study will compare monthly pregnancy testing to current practice in a double blind randomized control trial. As many women of childbearing age as possible will be recruited from the Hamilton Clinic for Opioid Substitutional Therapy. Women assigned to the intervention will have monthly testing at the same time as their monthly urine drug testing at the clinic. The primary objective is to assess if there is a significant difference is early pregnancy detection and the secondary objectives are to assess differences in pregnancy disposition and gestational age at entry to prenatal or abortion care.

DETAILED DESCRIPTION:
The Routine Pregnancy Screening in Women on Opioid Substitutional Therapy study involves screening women from the The Hamilton Clinic for OST regularly for pregnancy to determine if this results in earlier prenatal care and improved pregnancy disposition. All eligible women at the Hamilton clinic will be approached for recruitment. The study phase last for 18 months.

The investigators will assess for any significant difference in the rates of early pregnancy diagnosis, pregnancy disposition, and associated outcome measurements. Study results could inform best practices in the care of child-bearing women on OST and will provide baseline information and feasibility data to inform design of a larger RCT to assess the effect on pregnancy and birth outcomes.

This pilot study will serve to demonstrate whether routine pregnancy screening is effective for earlier pregnancy diagnosis and whether it has any impact on pregnancy disposition and entry into pregnancy-related care for women on OST. In addition, the investigators will also be seeking to address whether routine pregnancy testing is logistically and financially feasible for patients receiving OST at a primary care-run addiction setting. If this intervention is found to be both effective and feasible, it would be possible to apply this study methodology to larger-scale RCTs across multiple clinical sites with the power to assess maternal and fetal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* currently on methadone or buprenorphine maintenance therapy
* have some male sexual partners

Exclusion Criteria:

* females who have exclusively female sexual partners
* a previous diagnosis of premature menopause
* hysterectomy, oophorectomy, and/or tubal ligation
* current pregnancy
* current intrauterine device (hormonal or non-hormonal)
* unable to give informed consent in English

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Early Pregnancy Detection | 1.5 year
  Patients at the Hamilton Clinic present to the clinic most often on a weekly basis to provide a urine sample for urine drug screening and to meet with their MRP. This same urine sample can be tested for pregnancy in the intervention group once per month. Positive pregnancy test rates will be recorded for the intervention and control groups over the 1 year study period.

SECONDARY OUTCOMES:
Differences in pregnancy disposition | Through study completion, an average of 1.5 year
  Pregnancy disposition will be measured by the woman's choice to either continue with the pregnancy and enter care or enter into induced abortion care. Participants will either give the researchers access to their medical records and outcomes will be recorded from that information or participants can complete a self-report on pregnancy outcomes.
Gestational age at entry into pregnancy-related care | Through study completion, an average of 1.5 year
  Gestational age at entry into pregnancy related care will be obtained from ultrasounds and/or dates estimated from last menstrual period if access is granted to medical records. Otherwise researchers will depend on self-report. Pregnancy related care includes prenatal care or induced abortion services.
Cost of monthly pregnancy tests | 1.5 year
  The cost of additional pregnancy testing will be recorded by The Hamilton Clinic for OST for the length of the trial.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hamilton Clinic, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Heil SH, Jones HE, Arria A, Kaltenbach K, Coyle M, Fischer G, Stine S, Selby P, Martin PR. Unintended pregnancy in opioid-abusing women. J Subst Abuse Treat. 2011 Mar;40(2):199-202. doi: 10.1016/j.jsat.2010.08.011. Epub 2010 Oct 30. PMID 21036512
- [Background] Black AY, Guilbert E, Hassan F, Chatziheofilou I, Lowin J, Jeddi M, Filonenko A, Trussell J. The Cost of Unintended Pregnancies in Canada: Estimating Direct Cost, Role of Imperfect Adherence, and the Potential Impact of Increased Use of Long-Acting Reversible Contraceptives. J Obstet Gynaecol Can. 2015 Dec;37(12):1086-97. doi: 10.1016/s1701-2163(16)30074-3. PMID 26637081
- [Background] Armstrong KA, Kennedy MG, Kline A, Tunstall C. Reproductive health needs: comparing women at high, drug-related risk of HIV with a national sample. J Am Med Womens Assoc (1972). 1999 Spring;54(2):65-70, 78. PMID 10319594
- [Background] Sabourin JN, Burnett M. A review of therapeutic abortions and related areas of concern in Canada. J Obstet Gynaecol Can. 2012 Jun;34(6):532-542. doi: 10.1016/S1701-2163(16)35269-0. PMID 22673169
- [Background] Heaman MI, Newburn-Cook CV, Green CG, Elliott LJ, Helewa ME. Inadequate prenatal care and its association with adverse pregnancy outcomes: a comparison of indices. BMC Pregnancy Childbirth. 2008 May 1;8:15. doi: 10.1186/1471-2393-8-15. PMID 18452623
- [Background] Wong S, Ordean A, Kahan M; MATERNAL FETAL MEDICINE COMMITTEE; FAMILY PHYSICIANS ADVISORY COMMITTEE; MEDICO-LEGAL COMMITTEE; AD HOC REVIEWERS; SPECIAL CONTRIBUTORS. Substance use in pregnancy. J Obstet Gynaecol Can. 2011 Apr;33(4):367-384. doi: 10.1016/S1701-2163(16)34855-1. PMID 21501542